CLINICAL TRIAL: NCT03086616
Title: A Phase I and Early Efficacy Study of Convection Enhanced Delivery of Irinotecan Liposome Injection Using Real Time Imaging With Gadolinium in Children With Diffuse Intrinsic Pontine Glioma
Brief Title: CED With Irinotecan Liposome Injection Using Real Time Imaging in Children With Diffuse Intrinsic Pontine Glioma (DIPG) (PNOC 009)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sabine Mueller, MD, PhD (Other)
Collaborators: The V Foundation for Cancer Research (Other); Pacific Pediatric Neuro-Oncology Consortium (Other)
Responsible Party: Sponsor-Investigator, Sabine Mueller, MD, PhD, Associate Adjunct Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 160816; NCI-2017-01829 (Registry Identifier: Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2017-03-16; First posted 2017-03-22 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Diffuse Intrinsic Pontine Glioma
Keywords: DIPG; CED; glioma
MeSH Terms: conditions — Diffuse Intrinsic Pontine Glioma; Glioma | interventions — irinotecan sucrosofate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Newly Diagnosed DIPG (Experimental): Convection Enhanced Delivery (CED) of Nanoliposomal irinotecan (nal-IRI): Nal-IRI given directly into the tumor using a method called CED to newly diagnosed DIPG subjects after completion of radiotherapy. CED will be performed every 4-8 weeks. Drug concentration will start at 20mg/ml and escalate up to 40 mg/ml concentration.
  Interventions: Drug: Convection Enhanced Delivery (CED) of Nanoliposomal irinotecan (nal-IRI)

INTERVENTIONS:
Drug: Convection Enhanced Delivery (CED) of Nanoliposomal irinotecan (nal-IRI) — Nal-IRI will be given directly into the tumor using CED.
  Other Names: Irinotecan Liposome Injection

SUMMARY:
This is a Phase I and Early Efficacy Study of Convection Enhanced Delivery (CED) of irinotecan liposome injection (nal-IRI) Using Real Time Imaging with Gadolinium in Children with Diffuse Intrinsic Pontine Glioma who have completed focal radiotherapy

DETAILED DESCRIPTION:
This study will assess the safety and tolerability of repeated administration of nal-IRI co-infused with gadoteridol given by intratumoral CED in children with newly diagnosed DIPG.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed DIPG by MRI; defined as patients with a pontine location and diffuse involvement of at least 2/3 of the pons are eligible without histologic diagnosis. For lesions with typical imaging features, biopsy is neither encouraged nor required for eligibility. Tumors that are biopsied will be eligible if proven to be supportive of the diagnosis of a DIPG. Consensus of diagnosis by the study team must be met.
* Treatment must begin at a minimum of 4 weeks after, but no later than 14 weeks after, the date of the completion of focal radiotherapy.
* Prior Chemotherapy: Patients should be at least 30 days from last chemotherapy dose prior to start of CED infusion, with exception of antibody half-lives. For antibody therapies, at least 3 half-lives of the antibody after last dose of monoclonal antibody should have passed prior to CED infusion. Patients less than 30 days from last chemotherapy dose should be discussed with the study chair(s).
* Prior Radiation: Patients must have completed prior treatment with standard focal radiotherapy as part of initial treatment for DIPG and had their last dose at least 4 weeks prior to and no later than 14 weeks from the first CED treatment. Patients beyond 14 weeks from radiation therapy but with stable disease should be discussed with the study chair.
* Age ≥ 2 years of age. Patients younger than 3 years of age may be enrolled on study at the discretion of the Study Chair(s) if supporting evidence that brainstem lesion represents a brainstem glioma.
* Karnofsky ≥ 50 for patients > 16 years of age and Lansky ≥ 50 for patients 16 years of age and younger. Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
* Life expectancy of greater than 12 weeks measured from the date of completion of radiotherapy.
* Corticosteroids: Patients who are receiving dexamethasone must be on a stable or decreasing dose for at least 1 week prior to registration.
* Organ Function Requirements

  * Adequate Bone Marrow Function Defined as:Peripheral absolute neutrophil count (ANC) ≥1000/mm3 and platelet count ≥ 100,000/mm3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment) and normal coagulation defined as normal international normalized ratio (INR) or per institutional guidelines.
  * Adequate Renal Function Defined as:

    * Creatinine clearance or radioisotope glomerular filtration rate (GFR) ≥ 70 milliliters (mL)/min/1.73 m2 or
    * A serum creatinine based on age/gender as follows:

Age Maximum Serum Creatinine (mg/dL) Male Female 2 to < 6 years 0.8 0.8 6 to < 10 years 1 1 10 to < 13 years 1.2 1.2 13 to < 16 years 1.5 1.4

≥ 16 years 1.7 1.4

* Adequate Liver Function Defined as: Bilirubin (sum of conjugated + unconjugated) less than or equal to 1.5 x upper limit of normal (ULN) for age and serum glutamate pyruvate transaminase (SGPT) (ALT) less than or equal to 110 U/L. and Serum albumin ≥ 2 g/dL.
* Adequate Neurologic Function Defined as: Patients with seizure disorder may be enrolled if on non-enzyme inducing anticonvulsants and well controlled.

  * The effects of irinotecan liposome injection on the developing human fetus are unknown. For this reason women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation and 4 months after completion of irinotecan liposome injection administration. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
  * A legal parent/guardian or patient must be able to understand, and willing to sign, a written informed consent and assent document, as appropriate

Exclusion Criteria:

* Patients who had clinical and/or radiographic (MRI) progression of tumor following external beam radiation therapy.
* Patients with metastatic disease, including leptomeningeal or subarachnoid disseminated disease.
* Patients with tumor morphology or other imaging findings that predict poor coverage of the majority of the tumor including significant tumor volume outside the pons or presence of large cysts within the tumor that would prevent adequate tumor coverage by CED. Patients with concern for adequate tumor coverage based on tumor morphology should be discussed with the study chairs.
* Patients who are receiving any other tumor-directed therapy
* Patients with MRI or clinical evidence of uncontrolled tumor mass effect are excluded; the patients should be discussed with the study chair(s) and study neurosurgeon prior to any planned CED treatment.
* Untreated symptomatic hydrocephalus determined by treating physician.
* Patients should not be on enzyme-inducing anticonvulsants or other drugs that might interact with the cytochrome P450 enzyme system. If previously on an enzyme-inducing anti-epileptic drug (EIAED), patients should be off for at least 10 days prior to CED infusion and discussed with the Study Chair.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to irinotecan, topotecan, gadolinium, or lipids.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Female patients of childbearing potential must not be pregnant or breast-feeding. Female patients of childbearing potential must have a negative serum or urine pregnancy test within 14 days of registration.
* Patients who are unable to return for follow-up visits or obtain follow-up studies required to assess toxicity to therapy. Telemedicine visits are acceptable.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2021-10-04 (Actual); Study Completion 2021-10-04 (Actual)

PRIMARY OUTCOMES:
Number of Participants Experiencing Treatment-Related Adverse Events (AE) | 12 months
  Safety of repeated CED of nal-IRI following standard of care focal radiotherapy will be assessed by monitoring for adverse events, scheduled laboratory assessments, vital sign measurements, and physical examinations for subjects who receive the vaccination. The severity of toxicities will be graded according to the NCI CTCAE v4.0. Adverse events and clinically significant laboratory abnormalities (meeting Grade 3, 4, or 5 criteria according to CTCAE) will be summarized by maximum intensity and relationship to study drug(s). Grade 1 and 2 adverse events will be summarized if related to study therapy. Descriptive statistics will be utilized to display the data on toxicity

SECONDARY OUTCOMES:
Overall Survival (OS) at 12 months (OS12) | 12 months
  Any eligible subject treated on the dose level that will be investigated within the expansion cohort will be considered evaluable for clinical efficacy. Analyses will be performed after all enrolled patients have completed 12 months, or whenever the status of all patients has been established, whichever comes first. The primary analysis will be based on the Kaplan-Meier method. Kaplan-Meier estimates and the associated 95% confidence intervals (CI) will be calculated

OTHER OUTCOMES:
Distribution of Gadolinium | 12 months
  Assessment of observed distribution of gadolinium compared to pre-treatment modeling of the drug distribution utilizing predictive imaging software.

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Mueller, MD, PhD, MAS, Study Chair — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data after de-identification.
Supporting Information: Study Protocol